CLINICAL TRIAL: NCT03929978
Title: A Multi-Centre Post Market Clinical Follow-up Study Evaluating Performance and Safety of the SenSura® Mio Baby Device in Subjects With a Stoma
Brief Title: Performance and Safety Evaluation of the SenSura® Mio Baby Device in Subjects With a Stoma
Status: Withdrawn | Type: Observational
Why Stopped: lack of recruitment
Sponsor: Coloplast A/S (Industry)
Collaborators: Children's National Research Institute (Other); IWK Health Centre (Other); Driscoll Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CP280
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the non-interventional Post Market Clinical Follow-up (PMCF) study is to follow performance and safety of the newly marketed SenSura® Mio Baby device in a real-life setting.

The objective is to evaluate the SenSura® Mio Baby device performance and safety.

DETAILED DESCRIPTION:
The aim of the non-interventional Post Market Clinical Follow-up (PMCF) study is to confirm the established safety and performance of the newly marketed SenSura® Mio Baby device in a real-life setting.

The objective is to evaluate wear time of SenSura® Mio Baby device and other secondary endpoints related to performance, and safety of the device.

Primary endpoint:

• Median wear time

Secondary endpoints:

* Fulfillment of wear time expectations
* Number of unplanned change episodes
* Degree of leakage under the barrier
* Other areas of leakage
* Easiness of removal of barrier with Brava Baby Adhesive Remover
* Skin friendliness
* Evaluation of adhesive residues on skin after removal
* Frequency of refeeding
* Access for refeeding
* Hygienic refeeding procedure
* Frequency of pouch change
* Feeling of security
* Evaluation of SenSura® Mio Baby compared to Standard of Care (products used in the department) on comparative questions of performance (to be evaluated by nurses)
* Preference
* Number of adverse events

The study is a Post Market Clinical Follow-up Study, which is a descriptive study to confirm the established safety and performance of new ostomy devices recently device listed at the US market. Group 1 includes a retrospective data collection with the device used before the date of the study start. For Groups 2 and 3, data are not obtained for performance comparison to current ostomy device, but include prospective descriptive evaluations.

* Group 1: subjects having a stoma and using a Standard of Care device. These subjects will transfer to a SenSura® Mio Baby pouch
* Group 2: subjects who are newly operated. These subjects will be offered SenSura® Mio Baby pouch as their first device
* Group 3: subjects receiving medication such as chemotherapeutic treatment. These subjects may be newly operated subjects or already using a device. These subjects will transfer to a SenSura® Mio Baby pouch A total of 30 subjects needs to be enrolled in Group 1 and 2. A total of 6 subjects can be enrolled in Group 3.

For each Investigational site this means:

A total of 10 subjects needs to be enrolled in Group 1 and 2 and additional 2 subjects more can be enrolled in Group 3. However; the recruitment will be competitive between the 3 Investigational sites until the 30 subjects has been enrolled in Groups 1 and 2.

For details about the statistical analyses performed on this group of subjects, please see section 7.

At least 5 of the enrolled subjects should be in the age range from 30 Gestational Weeks (GW) up to 36 GW either from Group 1 or 2, in order to be able to confirm wear time and other performance related claims. In the primary evaluation, the mean median wear time will be compared to a threshold value of 24 hours which is based on a literature assessment of Standard of Care wear time performance.

Population The population in this study are (premature) infants over 30 weeks of gestation up to 6 months of age (cal-culated from term age meaning 40 GW) either with a colo- or, ileo-, or jejunostomy or a loop stoma, or two stomas placed closely together. Subjects can participate in the PMCF study if they fulfill the in-/exclusion criteria as listed in the tables below. However, the per protocol population include minimum 30 subjects from Group 1 or 2 as needed for the comparative performance evaluation.

Inclusion criteria To be included the subjects must: Justification

To ensure that:

1. Have a colostomy, ileostomy (jejunostomy), loop stoma, or two stomas placed closely together
2. Have given written informed consent (the legal authorized representative of the subject)

Exclusion criteria The subjects are not allowed to participate in case they: Justification

1) Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (assessed by the investigator)

The investigational device is SenSura® Mio Baby. SenSura® Mio Baby is a flat 2-piece (2P) ostomy device with an open bag and a baseplate, intended for premature infants over 30 weeks of gestation up to 6 months of age.

All devices in this study are approved for market release before study initiation.

Investigation approval

The non-interventional Post Market Clinical Follow-up (PMCF) study will be approved by local or central IRB in the US before study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria and justification hereof:

  1. Have a colostomy, ileostomy (jejunostomy), loop stoma, or two stomas placed closely together
  2. Have given written informed consent (the legal authorized representative of the subject)

Exclusion Criteria:

* The subjects are not allowed to participate in case they:

Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (assessed by the investigator)

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population in this study are (premature) infants over 30 weeks of gestation up to 6 months of age (calculated from term age meaning 40 GW) either with a colo- or, ileo-, or jejunostomy or a loop stoma, or two stomas placed closely together. Subjects can participate in the PMCF study if they fulfill the in-/exclusion criteria as listed in the tables below. However, the per protocol population include minimum 30 subjects from Group 1 or 2 as needed for the comparative performance evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Median wear time | 3 weeks